CLINICAL TRIAL: NCT04099589
Title: Multicenter Phase II Study of Gemcitabine/Cisplatin (GC) Chemotherapy Combined With PD-1 Inhibitor (Toripalimab) in the Neoadjuvant Treatment of Upper Urinary and Muscular Invasive Bladder Urothelial Carcinoma
Brief Title: Neoadjuvant Treatment of Upper Urinary and Muscular Invasive Bladder Urothelial Carcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Collaborators: Peking University First Hospital (Other); China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jianzhong Shou, Professor, Cancer Institute and Hospital, Chinese Academy of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC2121
Record Dates: First submitted 2019-09-19; First posted 2019-09-23 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Upper Tract Urinary Carcinoma; Muscle-invasive Bladder Cancer
Keywords: upper tract urinary carcinoma; muscle-invasive bladder cancer; neoadjuvant; chemotherapy; immunotherapy
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MIBC Group (Experimental): Muscle-invasive bladder cancer of T2-4aN0M0 confirmed by pathology after maximal transurethral resection of bladder tumors. Enrollment of 30 patients.
  Interventions: Drug: Toripalimab
- UTUC Group (Experimental): Upper tract urothelial carcinoma of T1-3N0M0 and high grade confirmed by flexible ureteroscope biopsy. Enrollment of 34 patients.
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Gemcitabine/Cisplatin plus Toripalimab

SUMMARY:
Few previous studies focused on the neoadjuvant treatments of upper urinary or bladder cancer, especially chemotherapy combined with immunotherapy, however, available data of retrospective studies showed this neoadjuvant treatment model might benefit patients. So This prospective Phase II clinical trial was designed to explore the efficacy of chemotherapy combined with PD-1 inhibitor as neoadjuvant therapy in upper urinary and muscle-invasive bladder urothelial carcinoma, then to improve the rate of complete pathological remission, survival and provide medical evidence.

ELIGIBILITY:
Inclusion Criteria:

1. bladder cancer of T2-4aN0M0
2. upper tract urinary carcinoma of T1-3N0M0 and high grade
3. ECOG 0-1
4. good organ function
5. no previous chemotherapy or immunotherapy
6. Informed consent form signed

Exclusion Criteria:

1. unable to receive chemotherapy or surgery due to physical abnormalities
2. previous cancer history
3. active tuberculosis
4. HIV
5. autoimmune disease
6. anticipating other clinical studies

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
pathological complete response rate | through study completion of 3 years
  the percentage of pT0N0 patients after operations

CONTACTS AND LOCATIONS:
Overall Officials: Jianzhong Shou, Principal Investigator — National Cancer Center/National Clinical Research Center for Cancer/Cancer Hospital, Chinese Academy of Medical Sciences and Peking Union Medical College
Locations (1):
- Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality, China